CLINICAL TRIAL: NCT01666847
Title: Milking the Umbilical Cord for Extreme Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Justin Josephsen M.D., Assistant Professor, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21429
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Infant, Extremely Premature
Keywords: Umbilical Cord Milking; Extremely Low Birth Weight Infant (ELBW)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cord Milking (Experimental): Infant receiving cord milking intervention before umbilical cord clamped.
  Interventions: Procedure: Milking the umbilical cord before cord clamping
- Immediate Cord Clamping (No Intervention): Infant whose umbilical cord is immediately clamped after delivery.

INTERVENTIONS:
Procedure: Milking the umbilical cord before cord clamping — The procedure will involve positioning the neonate below the level of the placenta and milking approximately 20cm of umbilical cord three times over 10-20 seconds total from the placental end to the neonate. The cord will then be clamped and the neonate handed to the awaiting medical team for routine care of a premature infant.
  Arms: Cord Milking

SUMMARY:
Milking the umbilical cord from the placental end toward the infant has been shown to benefit preterm infants when compared to either clamping the umbilical cord immediately or waiting delaying the clamping of the cord. Delaying cord clamping for 30-120 seconds has been shown to improve heart and lung function, reduces the need for blood transfusion, and reduces the risk for brain bleeding seen in some preterm infants. Delaying the clamping of the umbilical cord, however in extremely premature infants is not considered safe, since it also delays the resuscitation that these infants need immediately after birth. Milking the umbilical cord is believed have similar benefits to delaying the clamping of the cord, but can be done much faster (seconds rather than minutes). In this study, the cord will milked three times over about 10-20 seconds and the infant will be passed to the awaiting newborn medical team for routine care. Participants of this study will be randomly assigned to one of two study groups: the first group will have the cord milking intervention and the second group will not have any intervention other than routine, immediate cord clamping with routine care of mother and infant. Data will be collected about the mother prior to delivery and data will also be collected about the baby using computerized health records. The data will look at short term changes in red blood cell volumes, the need for blood transfusions, and rates of known complications of prematurity, including longer term developmental complications at 18-24 months.

The hypothesis is that milking the umbilical cord before cutting the cord will lead to a higher hemoglobin concentration and decrease the need for blood transfusions in extremely preterm neonates compared to the current standard of immediately clamping the umbilical cord.

DETAILED DESCRIPTION:
Eligible infants include singleton infants born between 24 and 27 6/7 weeks gestation who do not have congenital anomalies.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women/child pairs with infants born at an estimated gestation age between 24 0/7 and 27 6/7 weeks based on best estimate made by last menstrual period or ultrasound
* informed consent obtained by the pregnant women prior to delivery of the infant.

Exclusion Criteria:

* pregnancy with a multiple gestation
* infants with pre- or postnatally diagnosed major congenital anomalies or probable chromosomal abnormalities
* infants with hydrops fetalis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-10; Primary Completion 2016-08 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
To evaluate and compare hemoglobin and hematocrit concentrations in extremely low birth weight infants (ELVW) after cord milking intervention to ELBW infants receiving immediate cord clamping | Within 4 hour of birth
To evaluate and compare the incidence and numbers of blood transfusions after cord milking | Prior to initial infant discharge

SECONDARY OUTCOMES:
To evaluate and compare blood pressure after intervention and need for support medications | For first seven days of life
To evaluate and compare the incidence of hyperbilirubinemia and length of phototherapy | Three weeks
  Highest bilirubin or maximum at 120 hours of life, plus total days of phototherapy.
To evaluate the incidence of complications of prematurity in the study and control groups | Until 3 years corrected gestational age
To evaluate long term outcomes of prematurity in both groups in a follow-up study | Until 3 years corrected gestational age
To compare the difference in hemoglobin and hematocrit from umbilical cord blood | Within 4 hours of birth

CONTACTS AND LOCATIONS:
Overall Officials: Justin B Josephsen, MD, Principal Investigator — St. Louis University
Locations (2):
- United States (2):
  - Saint Louis University, Division of Neonatology, SSM Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Saint Louis University, Division of Neonatology, SSM St. Mary's Health Center, St Louis, Missouri

REFERENCES:
- [Background] Hosono S, Mugishima H, Fujita H, Hosono A, Minato M, Okada T, Takahashi S, Harada K. Umbilical cord milking reduces the need for red cell transfusions and improves neonatal adaptation in infants born at less than 29 weeks' gestation: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2008 Jan;93(1):F14-9. doi: 10.1136/adc.2006.108902. Epub 2007 Jan 18. PMID 17234653
- [Background] Leavitt BG, Huff DL, Bell LA, Thurnau GR. Placental drainage of fetal blood at cesarean delivery and feto maternal transfusion: a randomized controlled trial. Obstet Gynecol. 2007 Sep;110(3):608-11. doi: 10.1097/01.AOG.0000277262.80793.0d. PMID 17766607
- [Background] Rabe H, Jewison A, Fernandez Alvarez R, Crook D, Stilton D, Bradley R, Holden D; Brighton Perinatal Study Group. Milking compared with delayed cord clamping to increase placental transfusion in preterm neonates: a randomized controlled trial. Obstet Gynecol. 2011 Feb;117(2 Pt 1):205-211. doi: 10.1097/AOG.0b013e3181fe46ff. PMID 21252731
- [Background] Rabe H, Reynolds G, Diaz-Rossello J. Early versus delayed umbilical cord clamping in preterm infants. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD003248. doi: 10.1002/14651858.CD003248.pub2. PMID 15495045
- [Background] Rabe H, Reynolds G, Diaz-Rossello J. A systematic review and meta-analysis of a brief delay in clamping the umbilical cord of preterm infants. Neonatology. 2008;93(2):138-44. doi: 10.1159/000108764. Epub 2007 Sep 21. PMID 17890882